CLINICAL TRIAL: NCT03765125
Title: Dietary Intake of Collagen Peptides and Its Effects on Periodontal Inflammation - a Randomized Clinical Trial
Brief Title: Dietary Collagen Peptides and Periodontal Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VERIPA17
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2019-04

CONDITIONS: Gingivitis
Keywords: gingivitis; collagen peptide; plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled 2-arm, parallel group
Who Masked: Participant, Investigator
Masking Description: test and placebo powder contained in coded blister packages of identical shape and colour Handing out of the assigned powder by a study nurse not involved in the clinical examination and data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- collagen peptide test (Experimental): 1 x daily consumption of 1 blister package of the collagen-peptide test powder dissolved in water over a period of 90 days
  Interventions: Dietary Supplement: collagen peptide test
- collagen peptide placebo (Placebo Comparator): 1y daily consumption of 1 blister package of the placebo powder dissolved in water over a period of 90 days
  Interventions: Dietary Supplement: collagen peptide placebo

INTERVENTIONS:
Dietary Supplement: collagen peptide test — Collagen peptides from bovine skin with an average molecular weight of approx. 2,000 g/mol. Average particle size is about 150 μm.
  Other Names: collagen peptide placebo
  Arms: collagen peptide test
Dietary Supplement: collagen peptide placebo — collagen peptide placebo
  Arms: collagen peptide placebo

SUMMARY:
This randomized, double-blind, placebo-controlled 2-arm, parallel group clinical trial is designed to evaluate the impact of the regular consumption of collagen peptides on the clinical signs of gingival and periodontal inflammation in a cohort of patients suffering from periodontal disease.

DETAILED DESCRIPTION:
The positive influence of the regular consumption of bioactive collagen peptides on connective tissue and skin physiology has already been documented by several clinical trials. Preliminary data of an observational clinical trial involving periodontitis patients suggest that the adjunctive consumption of bio-active collagen peptides may also improve the outcome of established periodontitis therapy comprising the professional mechanical removal of disease-associated bacterial biofilms from exposed root surfaces.

This randomized, double-blind, placebo-controlled 2-arm, parallel group clinical trial is designed to evaluate the impact of the regular, 3-month consumption of collagen peptides on clinical and microbiological parameter of periodontal health in a cohort of periodontal recall patients with the following endpoints:

Primary Endpoint:

Change in the percentage of periodontal pockets being positive for bleeding on probing (BoP) after the consumption of the collagen peptides in comparison to the consumption of a placebo product

Secondary Endpoints:

1. changes in probing pocket depth (PPD)
2. changes in clinical attachment level (CAL)
3. changes in the periodontal inflammatory load as assessed by the calculation of the periodontal inflamed surface area (PISA) index
4. changes in Gingival Index (GI) scores
5. changes in Plaque Control Record (PCR) scores
6. changes in Plaque Index scores
7. changes in the composition of the sulcular/pocket microbiota
8. changes in the composition of the intestinal microbiota

Examiner calibration is performed before the onset of the trial and is repeated in 8 weeks intervals throughout the trial.

Sample Size Calculation As this is the first controlled clinical trial evaluating the impact of collagen peptide consumption on the extent of periodontal inflammation, sample size calculation is based on substitute data from preceding studies demonstrating an increase in tissue healing by up to 30%.

With a given difference of 30% reduction in the number of bleeding periodontal pockets (BoP) and an assumed standard deviation of 30% , sample size calculation resulted in a minimum of 19 subjects per group in order to be able to statistically verify differences with a power of 80%, and p<0.05.

Chi-square-test with maximum likelihood method will be used for the analysis of categorical variables, Mann-Whitney U-test will be used for the analysis of independent samples, and Wilcoxon signed rank test for the analysis of paired samples. The level of significance will be set to p≤0.05.

Study patients will be recruited from periodontitis patients seeking routine periodontal maintenance care comprising professional mechanical plaque removal (PMPR) at the Dept. of Periodontology of the University Hospital Wuerzburg.

At baseline prior to the performance of PMPR all above-mentioned study parameters will be recorded. Subsequently the study participants will be randomly assigned to the experimental groups (test/placebo) and a supply of the assigned product (test/placebo) will be given to them with the instruction to consume it 1 x daily for the 3-month duration of the trial.

At 2 months (visit 2) and at 3 months (end of study) after the baseline examination all clinical and microbiological parameters will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* number of teeth ≥ 10
* age ≥ 35 ≤ 70 years
* body mass index (BMI) ≥ 24 ≤ 30
* history of periodontal disease and inclusion in a regular scheme of supportive periodontal therapy (regularly repeated subgingival biofilm removal 2-4 x/year)
* presence of mild to moderate gingivitis (Gingiva Index > category GI 0 ≤ category GI 2) at a minimum of 3 teeth

Exclusion Criteria:

* manifestation of inflammatory oral mucosal diseases other than gingivitis
* xerostomia (salivary flow ≤ 0.1 ml/minute)
* inability for regular oral home care
* inability to follow the study protocol due to intellectual or physical handicaps
* history of malignancy, radiotherapy, or chemotherapy for malignancy in the past 5 years
* current pregnancy
* acute infections as HIV
* existence of metabolic bone disease
* smoking status of more than 10 cigarettes/day
* use of antibiotics and/or anti-inflammatory medication within 4 weeks prior to screening.
* active orthodontic therapy
* diabetes mellitus type I and II
* regular consumption of medications interfering with gingival inflammation (e.g. cortisol)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of periodontal sites being positive for bleeding on probing (BoP) | 90 days
  Bleeding on probing will be recorded at 6 sites per tooth after gentle probing of the periodontal sulcus/pocket.

SECONDARY OUTCOMES:
clinical attachment level (CAL) | 90 days
  clinical attachment level will be assessed using a manual periodontal probe
pocket probing depth (PPD) | 90 days
  pocket depth will be assessed using a manual periodontal probe
periodontal inflamed surface area (PISA) | 90 days
  PISA values will be calculated using the recorded BoP, CAL and PPD data
modified Gingival Index | 90 days
  The modified Gingival Index will be recorded from the buccal aspect of all teeth
Plaque Control Record | 90 days
  The extension of plaque along the gingival margin will be assessed from the mesial, distal, buccal and oral aspects of all teeth using a standard periodontal probe.
Plaque Index | 90 days
  The Plaque Index will be recorded from the vestibular aspects of the teeth 16, 21, 24, 36, 41, 44
Composition of the oral microbiota | 90 days
  Subgingival plaque samples will be collected by paper points from the 4 deepest periodontal pockets of each patient and subsequently analysed by whole genome sequencing
Composition of the intestinal microbiota | 90 days
  Stool samples will be collected from each study participant and subsequently analysed by whole genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Jockel-Schneider, Dr., Principal Investigator — Wuerzburg University Hospital
Locations (2):
- Germany (2):
  - Dept. of Periodontology, University Hospital Wuerzburg, Würzburg
  - Section of Periodontology, Würzburg

IPD SHARING:
Plan to Share IPD: No